CLINICAL TRIAL: NCT03703596
Title: Efficacy and Safety of Anlotinib Versus Docetaxel in Advanved Non-squamous Non-small-cell Lung Cancer Without EGFR Mutation Who Failed in First-line Platinum-based Doublet Chemotherapy: an Open, Muti-center, Randomized Controlled Trial
Brief Title: Anlotinib Versus Docetaxel as the Second-line Treatment in EGFR Wild Type Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jianing Tang, assistant of Medical Oncology Thoracic Department, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L023
Record Dates: First submitted 2018-09-19; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Lung Cancer; Lung Cancer Metastatic
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib hydrochloric (Experimental): Anlotinib (12mg QD PO d1-14, 21 days per cycle)
  Interventions: Drug: Anlotinib Hydrochloride
- Docetaxel (Experimental): Docetaxel (75mg/m2 IV d1, 21 days per cycle)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib (12mg QD PO d1-14, 21 days per cycle)
  Arms: Anlotinib hydrochloric
Drug: Docetaxel — Docetaxel (75mg/m2 IV d1, 21 days per cycle)
  Arms: Docetaxel

SUMMARY:
This study is conducted to explore the safety and efficacy of anlotinib, a tyrosine kinase inhibitors of Vascular Endothelial Growth Factor Receptor 2（VEGFR）、FGFR（Fibroblast Growth Factor Receptor）, Platelet-derived growth factor Receptor（PDGFR） and c-kit, vs docetaxel in advanced Non-squamous Non-small cell lung cancer harbouring wild-type epidermal growth factor receptor (EGFR) .

DETAILED DESCRIPTION:
This is a multicentre randomised controlled clinical trial conducted in China to compare the efficacy and and safety of Anlotinib vs Docetaxel in patients of EGFR mutation-negative advanced nonsquamous non-small Cell Lung Cancer.

Eligible patients will be randomized to arm A and arm B:

Arm A: Patients on the anlotinib arm received 12mg anlotinib orally daily on day 1 to 14 of a 21-day cycle.

Arm B: Patients on the docetaxel arm received 75mg/m2 docetaxel as intravenous infusion on day 1 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* -≥ 18 and ≤ 70 years of age. Signed the informed consent form prior to patient entry
* Histologically or pathologically confirmed non-squamous non-small cell lung cancer(NSCLC) with stage IV .
* Histologically or pathologically confirmed non-squamous non-small cell lung cancer(NSCLC) with stage IV .
* Patients who has failed from the first-line Platinum-based Doublet chemotherapy harbouring epidermal growth factor receptor(EGFR) sensitive mutations negetive, confirmed by pathological or blood test results) ）,ALK/ROS1 mutation-negative or unknown (For recurrent patients, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant were assessed for eligibility, and the last treatment time must be more than 6 months before enrollment） Noted: failed from prior treatment means(1) progress disease confirmed by CT; cannot tolerable from standard treatment, such as hematologic toxicities ≥ level 4; non-hematologic toxicities ≥ level 3;damages of heart/liver/kidney ≥ level 2 in CTC AE 4.0
* Must have at least one measurable lesion as per RECIST 1.1 defined as a lesion that is 10mm in longest diameter imaged by CT scan or MRI；prior topical treatment, such as radiotherapy cryosurgery to the lesions is not allowed in less than 3 months;
* Life expectancy ≥3 months.
* Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
* Toxicity caused by prior anti-cancer treatments was restored to ≤ level 1 in CTC AE (4.0) , except alopecia;
* The blood routine examination need to be standard (no blood transfusion and blood products within 14 days, no g-csf and other hematopoietic stimulating factor correction); Hemoglobin（HB）≥90 g/L; A Neutrophil count of （ANC）≥1.5×10e9/L; A Platelet count of （PLT）≥80×10e9/L; A Total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL); A alanine aminotransferase (ALT) and a aspartate aminotransferase (AST) of ≤2.5 UNL, in case of liver metastasis ALAT and ASAT≤5 UNL; A creatinine (Cr) of ≤1.5 UNL; a creatinine clearance rate ≥ 60ml/min (Cockcroft-Gault);
* The woman patients of childbearing age who must agree to take contraceptive methods during the research and within another 8 weeks after it and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; the man patients who must agree to take contraceptive methods during the research and within another 8 weeks Voluntarily joined the study and signed informed consent, with good compliance and follow-up.

Exclusion Criteria:

* -Mixed Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer, adenocarcinoma mixed with squamous cell carcinoma
* No squamous NSCLC with hemoptysis (>50ml/day);
* Treated by taxel or similar drugs in 12months;
* symptoms of brain metastases cannot be controlled and treated within less than 2 months
* Tumor locate within a distance of less than 5 mm from the large vessels, less than 2 cm from the bronchial tree, or has invaded local large vessels; tumor with cavum or necrotic obviously;
* Uncontrolled hypertension (systolic ≥140mmHg and/or diastolic ≥90mmHg, despite optimal drug therapy).
* Patients with with grade Ⅱ myocardial ischemia or myocardial infarction, poor control of arrhythmias (including QTc interval male ≥ 450 ms, female ≥470 ms); according to NYHA standard, grade Ⅲ ~ Ⅳ heart failure, or cardiac color Doppler ultrasound examination showed left ventricular ejection fraction (LVEF) <50%.
* Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment;note: Note: under the premise of International Normalized ratio (INR) of prothrombin time (PT) Less than or equal to 1.5, allow to administrate low-dose heparin (adult daily dose is 06000 ~ 12000 U) or low-dose aspirin (100 mg daily dosage or less) , for prophylactic purposes
* Patients whose routine urine tests indicate that urine protein ≥ ++ or verifies that the 24-h urine protein quantitation ≥ 1.0 g.
* Patients whose has peripheral neuropathy over level 2 in CTC AE4.0, except trauma.
* Patients with respiratory syndrome (difficulty breathing of level 2 or higher ), serous cavity effusion need to surgical treatment ( including pleural of level 2 or higher with respiratory distress and anoxia
* Patients who have unhealed wounds or fractures for a long time.
* Patients with severe infections , and need to receive systemic antibiotic treatment
* Decompensated diabetes or other contraindication with high dose glucocorticoid therapy;
* Cirrhosis or decompensated liver disease; active or untreated hepatitis C and/or Hepatitis B virus (HBV) infection（prior hepatitis B history, HBsAg positive and HBV DNA≥500IU/mL; HCV RNA positive and hepatic Insufficiency
* Has an obvious factor influencing oral drug absorption, such as unable to swallow, chronic diarrhea and intestinal obstruction, etc
* Patients who received major surgical operations or experienced severe traumatic injuries, bone fracture, or ulcers within 4 weeks before screening.
* Severe weight loss (> 10%) Within 6 weeks before Random
* Patients who had obvious hemoptysis (>50ml/day) within 3 months before screening; Patients who experienced bleeding symptoms of clinical significance within 3 months before screening, or with confirmed bleeding tendency such as hemorrhage of digestive tract, hemorrhagic gastric ulcer, baseline occult blood in stool ++ and above, or vasculitis, etc;
* Patients who manifested arterial/venous thrombus events, e.g. cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, etc., within 12 months before screening.
* Allergic reactions to anotol or excipients in experimental drugs.
* Allergic reactions to contrast medium
* Patients have participated in other antitumor drug clinical trials Within 4 weeks before enrollment or prepare to receive systemic anti-tumor treatment during the study or Within 4 weeks before randomization
* Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-10-16 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to 24 months
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.
Disease Control Rate (DCR) | Up to 24 months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Wenxiu Yao, PhD, Principal Investigator — Director of Medical Oncology Thoracic Department
Locations (10):
- China (10):
  - People's hospital of deyang city, Deyang, Sichuan
  - Chengdu fifth people's hospital, Chengdu
  - Sichuan cancer hospital, Chengdu
  - People's hospital of guangan city, Guangan
  - The affiliated hospital of southwest medical university, Luzhou
  - Nanchong central hospital, Nanchong
  - Neijing second people's hospital, Neijiang
  - Suning central hospital, Suning
  - Zigong first people's hospital, Zigong
  - Zigong fourth people's hospital, Zigong

IPD SHARING:
Plan to Share IPD: No